CLINICAL TRIAL: NCT06873815
Title: A Single-Arm Prospective Trial of Fluorescein Mapping in Patients Undergoing Vulvectomy for Extramammary Paget's Disease
Brief Title: A Study of Fluorescein Sodium in People Undergoing Vulvectomy for Extramammary Paget's Disease (EMPD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-002
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Extramammary Paget's Disease
Keywords: Fluorescein Mapping; Vulvectomy; 25-002
MeSH Terms: conditions — Paget Disease, Extramammary | interventions — Fluorescein

STUDY DESIGN:
Intervention Model Description: This is a prospective single-arm intervention study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Undergoing Vulvectomy for Extramammary Paget's Disease (EMPD) (Experimental): Consented patients will receive IV fluorescein sodium in the operating room before the vulvectomy procedure.
  Interventions: Drug: Fluorescein Sodium

INTERVENTIONS:
Drug: Fluorescein Sodium — Patients will receive IV fluorescein sodium in the operating room before the vulvectomy procedure.

SUMMARY:
The researchers are doing this study to see if giving people fluorescein sodium as an IV infusion before their vulvectomy for treating extramammary Paget's disease (EMPD) can help surgeons with performing the procedure. The researchers will look at whether fluorescein sodium helps surgeons identify disease cells that should be removed. Other purposes of this study include looking at the following: If there are any complications during or after vulvectomy involving the use of fluorescein sodium. If fluorescein sodium can reveal tissue that surgeons cannot operate on (unresectable tissue).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Noninvasive or microinvasive EMPD with a contiguous visible clinical lesion
* Newly diagnosed or recurrent lesion
* Scheduled to undergo wide local excision or vulvectomy not requiring resection of the clitoris, urethra, or anus and with the surgeon's judgment that primary closure is possible (V-Y advancement flap closure is allowed)

Exclusion Criteria:

* History of allergic reaction to fluorescein sodium
* Multifocal, noncontiguous clinical lesion
* Current or previous invasive EMPD
* History of invasive vulvar, vaginal, or anal cancer
* Lesion in which resection of the clitoris, urethra, and/or anus is deemed to be necessary
* Lesion in which a primary closure or V-Y advancement flap is believed not to be possible and a larger myocutaneous flap is needed for closure of the defect
* History of radiation therapy to the vulva and/or anus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — People Undergoing Vulvectomy for Extramammary Paget's Disease (EMPD)
Enrollment: 27 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
rate of positive pathologic surgical margin status | 1 year
  is to determine whether the use of IV fluorescein sodium reduces the rate of positive surgical margins in patients undergoing vulvectomy for EMPD. The incidence of positive surgical margins on final pathology will be evaluated as the primary endpoint;

SECONDARY OUTCOMES:
incidence of intraoperative or postoperative complications | up to 30 days post op
  all intraoperative and postoperative complications (including allergic reactions to fluorescein sodium injection, allergic reaction, infection, wound breakdown, need for reoperation) in the study population will be recorded prospectively. All complications of grade 3 or higher, as defined by Martin et al.10

CONTACTS AND LOCATIONS:
Overall Officials: Mario Leitao, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm